CLINICAL TRIAL: NCT03893396
Title: Safety Assessment of Angioplasty Procedures
Acronym: SCRAP
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier de la Rochelle Ré Aunis (Other)
Collaborators: BBraun Medical SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018/P02/283
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Angiospastic; Disorder
Keywords: drug eluting stent; Drug-coated balloon; Bare-Metal Stent; Revascularization
MeSH Terms: interventions — Angioplasty, Balloon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Coronary angioplasty — Procedure used to open clogged heart arteries. Involves the insertion of a tiny balloon and/or a stent to widen the artery.
  Other Names: Percutaneous coronary

SUMMARY:
Ischemic heart disease, or coronary heart disease, covers a set of pathologies due to insufficient oxygen supply to the myocardium due to the development of atherosclerosis in one or more coronary arteries. To evaluate the safety of angioplasty performed in patients operated on at La Rochelle Hospital, the rate of major adverse cardiac events (MACE) will be determined and compared with data from the literature.

DETAILED DESCRIPTION:
The use of active stents for the treatment of coronary stenosis is currently the standard treatment in almost all types of coronary lesions. In percutaneous transluminal treatment of coronary lesions, balloon angioplasty and bare stents have not shown satisfactory results in the past. The so-called active drug-eluting balloon could represent a new therapeutic option for the treatment of de novo lesions.

ELIGIBILITY:
Inclusion Criteria:

* Interventional revascularization of a coronary lesion,
* Member or beneficiary of a social security system,
* Informed of the study.

Exclusion Criteria:

* Language barrier,
* Minor,
* Pregnant woman,
* Person under guardianship,
* Person deprived of his/her liberty,
* Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for coronary angiography for revascularization are those for whom a diagnosis of acute (Acute Coronary Syndrome with or without ST segment elevation) or chronic (Silent myocardial ischemia, angina) coronary pathology has been made
Sampling Method: Non-Probability Sample
Enrollment: 983 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ludovic MEUNIER, MD, Study Director — Groupe Hospitalier de la Rochelle Ré Aunis
Locations (1):
- Groupe Hospitalier de la Rochelle Ré Aunis, La Rochelle, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available with publication. A Digital Object Identifier will be used.
  Keywords are Coronary Artery Disease, Percutaneous Coronary Intervention, Angioplasty, Drug-eluting stent, Drug-coated balloon, Patient Outcome Assessment.
  The only available version will be the locked database. With the exception of dates, all data will be made available. Dates will only be collected to verify the quality of the clinical trial execution. They do not add to the clinical question, and may be a means of indirectly identifying patients. The database will be made available through Zenodo.
  Medical Subject Headings (MESH) terms will be used to describe clinical data. International standard unit will be used. The data will be made available to the community of scientists and clinicians interested in percutaneous coronary intervention.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available with the free access to the publication for 15 years.
Access Criteria: A Digital Object Identifier will be provided
URL: https://doi.org/10.5281/zenodo.8182420

REFERENCES:
- [Result] Meunier L, Godin M, Souteyrand G, Mottin B, Valy Y, Lordet V, Benoit C, Bakdi R, Laurencon V, Genereux P, Waliszewski M, Allix-Beguec C. Prospective, single-centre evaluation of the safety and efficacy of percutaneous coronary interventions following a decision tree proposing a no-stent strategy in stable patients with coronary artery disease (SCRAP study). Clin Res Cardiol. 2023 Sep;112(9):1164-1174. doi: 10.1007/s00392-022-02054-7. Epub 2022 Jul 1. PMID 35776144
- [Derived] Meunier L, Eccleshall S, Bakdi R, Godin M, Souteyrand G, Mottin B, Valy Y, Benoit C, Lordet V, Laurencon V, Milhem A, Waliszewski M, Allix-Beguec C. Long-Term Effectiveness of a Stent-Less Strategy With Drug Coated Balloon in Coronary Artery Disease: 3-Year Follow-Up of a Prospective All-Comers Observational Study. Clin Cardiol. 2025 Aug;48(8):e70189. doi: 10.1002/clc.70189. PMID 40745698

RESULTS

PARTICIPANT FLOW:
Groups:
- c-DES: If the patient was hemodynamically or rhythmically unstable, conventional drug-eluting stent (DES) angioplasty was performed
- BO-DES: Patients eligible for a stent-less strategy underwent lesion preparation with scoring balloon. In cases of persistent residual stenosis, dissection at high risk of acute occlusion, or dissection at risk of secondary aneurysmal, bailout stenting with DES was performed (BO-DES)
- DCB-only: Patients eligible for a stent-less strategy underwent lesion preparation with scoring balloon. If lesion preparation was successful, the second step of angioplasty was performed with drug-coated balloon (DCB).
Period: Overall Study
Arm/Group | c-DES | BO-DES | DCB-only
Started | 143 | 294 | 546
One-year Follow-up | 138 | 281 | 530
Completed | 127 | 268 | 501
Not Completed | 16 | 26 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | c-DES | BO-DES | DCB-only | Total
Number analyzed (Participants) | 143 | 294 | 546 | 983
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (13.5) | 69.0 (11.4) | 68.4 (11.3) | 68.6 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 72 | 137 | 250
  Male | 102 | 222 | 409 | 733
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 143 | 294 | 546 | 983
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 27.3 (4.5) | 27.4 (4.4) | 27.4 (5.0) | 27.4 (4.7)
Clinical presentation [Count of Participants; unit: Participants]
  ST-elevation myocardial infarction (STEMI) | 58 | 54 | 61 | 173
  Non-ST-Elevation Myocardial Infarction (NSTEMI) | 37 | 87 | 120 | 244
  Chronic coronary syndrome | 48 | 153 | 365 | 566

OUTCOME MEASURES:

1. Primary Outcome: Number of Major Adverse Cardiac Events (MACE)
Description: The primary endpoint is a composite endpoint that includes major adverse cardiac events defined as cardiovascular death, non-fatal myocardial infarction (MI), non-fatal stroke (stroke) and revascularization of target lesion (TLR) within 12 months of surgery.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- DCB-only: Patients eligible for a stent-less strategy underwent lesion preparation with scoring balloon. If lesion preparation was successful, the second step of angioplasty was performed with DCB.
Arm/Group | c-DES | BO-DES | DCB-only
Number analyzed (Participants) | 138 | 281 | 530
Participants
  Number of in-hospital death following percutaneous coronary intervention | 9 | 6 | 2
  Number of participants without MACE | 119 | 254 | 509
  Number of participants who underwent MACE | 10 | 21 | 19

2. Secondary Outcome: Number of Major Adverse Cardiac Events (MACE)
Description: The secondary endpoint is a composite endpoint that includes major adverse cardiac events defined as cardiovascular death, non-fatal myocardial infarction (MI), non-fatal stroke (stroke) and revascularization of target lesion (TLR) within 12 months of surgery.
Time Frame: 36 months
Population: All consecutive patients in whom coronary angioplasty was performed, i.e. acute coronary syndrome non-ST myocardial infarction (NSTEMI) or ST myocardial infarction (STEMI), chronic coronary syndrome including angina, silent ischemia, ischemic heart disease, were eligible. The exclusion criteria were patients <18 years of age, pregnancy, legally protected patients or deprived of liberty, and refusal to participate. In-hospital deaths following percutaneous coronary intervention were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | c-DES | BO-DES | DCB-only
Number analyzed (Participants) | 118 | 262 | 499
Participants
  Number of participants without MACE | 94 | 218 | 438
  Number of participants who underwent MACE | 24 | 44 | 61

ADVERSE EVENTS:
Time Frame: Up to three year after percutaneous coronary intervention
Arm/Group | c-DES | BO-DES | DCB-only
All-Cause Mortality (participants affected / at risk) | 26/143 | 31/294 | 43/546
Serious Adverse Events (participants affected / at risk) | 9/143 | 19/294 | 22/546
Other Adverse Events (participants affected / at risk) | 0/143 | 0/294 | 0/546
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | c-DES (N=143) | BO-DES (N=294) | DCB-only (N=546)
Coronary restenosis (Cardiac disorders) | 4 (5) | 16 (19) | 13 (15)
Stroke (Nervous system disorders) | 4 (4) | 2 (2) | 6 (6)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT03893396/Prot_SAP_000.pdf